CLINICAL TRIAL: NCT03431766
Title: A Prospective, Randomized-controlled Study of the Effect of a Chlorhexidine Based Gel on the Internal Implant Surface Treatment on the Reduction of Bacterial Load and on the Regressive Bone Modelling.
Brief Title: 0.2% Chx Gel vs Implant Bacterial Contamination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, full time professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2342
Record Dates: First submitted 2018-01-15; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Bone Resorption; Bacteria Caused Disease
Keywords: chlorhexidine gel; dental implant
MeSH Terms: conditions — Bone Resorption; Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group A (Placebo Comparator): on this group a placebo gel will be applied on the internal surface of the implant during all the surgical and prosthetic phases of the treatment.
  Interventions: Device: placebo gel
- test group B (Experimental): on this group a 0.20% chlorhexidine gel will be applied on the internal surface of the implant during all the surgical and prosthetic phases of the treatment described on the study protocol.
  Interventions: Device: 0.20% chlorhexidine gel

INTERVENTIONS:
Device: placebo gel — On control group A once the dental implants are inserted on both mandible or maxilla of the patient placebo (group A) would be applied on the internal surface of the implants on all the surgical or prosthetic phases of the study.
  Arms: control group A
Device: 0.20% chlorhexidine gel — On test group B once the dental implants are inserted on both mandible or maxilla of the patient a 0.20% chlorhexidine gel would be applied on the internal surface of the implants on all the surgical or prosthetic phases of the study.
  Arms: test group B

SUMMARY:
The objective of this human randomized, double blind, placebo-control (RDBPC) study is to evaluate the efficacy of a 0.2% chlorhexidine (CHX) gel on reducing bacterial load and peri-implant inflammation at implant-abutment interface during the early healing stage.Thirty-six healthy patients (mean age 52,28 years; range 29-75 years) without a significant past medical anamnesis, all non-smokers, will be recruited as candidates for single implant placement and prosthetic rehabilitation.Patients will be randomly divided in group A (control) and group B (test) as indicated by the randomization chart. All Implants (Cortex classic, Shalomi, Israel)would be inserted by two skilled operators who followed a two-stage protocol and placed them according to the manufacturer's instructions.Eventually, all patients will be rehabilitated with a single implant-supported crown. During all the stages either a gel containing 0.20% CHX (Plak ®Gel; Polifarma Wellness Srl, Rome, Italy) or a placebo gel (Placebo, Polifarma Wellness Srl, Rome, Italy) will be used. The two gels are perfectly alike in packaging, color and smell and nobody knew the exact location of placebo or test gel, which will be revealed, only after data collection would be performed, by the person who prepared them. A or B gel will be placed on the internal connection abutments and then a cover screw would be inserted. Finally, the site would be sutured with non-absorbable nylon sutures. Cone Beam Computed Tomography evaluation (CBCT) (VatechIpax 3D PCH-6500, Fort Lee, NJ USA) would be performed both for pre-operative and post-surgical implant placement. Both gels will be given to the patients, according to the protocol, and applied 2 times/day until suture removal after 7 days. Soft tissue biopsies would be performed by means of a circular scalpel (5.5 mm in diameter) at the implant insertion (T0) and after two months of healing (second stage surgery)(T1) to analyze the peri-implant inflammatory infiltrate and the micro-vessel density (MVD) in both groups. All the radiographs taken during the study time points would be analysed to measure the bone resorption after 1 year or on other studt time points.

DETAILED DESCRIPTION:
The objective of this human randomized, double blind, placebo-control (RDBPC) study is to evaluate the efficacy of a 0.2% chlorhexidine (CHX) gel on reducing bacterial load and peri-implant inflammation at implant-abutment interface during the early healing stage. Thirty-six healthy patients (mean age 52,28 years; range 29-75 years) without a significant past medical anamnesis, all non-smokers, will be recruited as candidates for single implant placement and prosthetic rehabilitation.Patients will be randomly divided in group A (control) and group B (test) as indicated by the randomization chart. The randomization of this prospective, randomized-controlled, double blind study was obtained using computer generated random numbers, centralized with sequentially sealed opaque envelopes provided by the study adviser.The surgeon will open the sealed envelope containing the randomized group only after having inserted the implant.During the first evaluation, all subjects will be clinically examined: radiographs, plaque and bleeding scores would be carried out for diagnostic evaluation; then the patients would be scheduled for surgery procedures. All Implants (Cortex classic, Shalomi, Israel) would be inserted by two skilled operators who will follow a two-stage protocol and would place them according to the manufacturer's instructions. Before surgery all the patients would be subject to applications of chlorhexidine digluconate solution 0.2% for 2 minutes to obtain lower bacterial load and local anesthesia would be given with Articaine® (Ubistesin 4% - Espe Dental AG Seefeld, Germany) associated with epinephrine (1:100.000). Eventually, all patients would be rehabilitated with a single implant-supported crown. During all the stages either a gel containing 0.20% CHX (Plak ®Gel; Polifarma Wellness Srl, Rome, Italy) or a placebo gel (Placebo, Polifarma Wellness Srl, Rome, Italy) would be used. The two gels are perfectly alike in packaging, colour and smell and nobody knows the exact location of placebo or test gel, which would be revealed, only after data collection would be performed, by the person who prepared them. A or B gel would be placed on the internal connection abutments and then a cover screw would be inserted. Finally, the site would be sutured with non-absorbable nylon sutures. Cone Beam Computed Tomography evaluation (CBCT) (VatechIpax 3D PCH-6500, Fort Lee, NJ USA) would be performed both for pre-operative and post-surgical implant placement. All patients will recieve antibiotic therapy, 2g/day for 6 days (Augumentin®; Glaxo-Smithkline Beecham, Brentford, UK).The post-operative pain would be controlled with NSAIDs, and oral hygiene instructions would be given. Both gels would be given to the patients, according to the protocol, and applied 2 times/day until suture removal after 7 days. Soft tissue biopsies would be performed by means of a circular scalpel (5.5 mm in diameter) at the implant insertion (T0) and after two months of healing (second stage surgery)(T1) to analyze the peri-implant inflammatory infiltrate and the micro-vessel density (MVD) in both groups.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sex between 18 and 75 years,
* good systemic and oral health,
* need of single crown implant supported restoration,
* at least six months of healing after tooth extraction,
* cortical bone thickness > 5 mm measured by means of a cone beam computed tomography (CBCT).

Exclusion Criteria:

* poor oral hygiene,
* active periodontal disease or other oral disorders,
* insufficient bone thickness for implant insertion,
* bone augmentation procedures,
* immediate loading protocols,
* uncontrolled diabetes mellitus,
* immune diseases,
* smoking
* bruxism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-11-17 (Actual); Primary Completion 2019-01-12 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
bone resorption around dental implants on both study groups | 1 year after implant placement
  The bone resorption will be measured on periapical radiographs that would be taken during the clinical phases of the study. It would be used also an individual bite block to assure the reproducibility of the same position during all the phases. The distance between the crestal bone level and the first point where the bone attaches to the implant will be measured. The measurements will be in millimetres.

SECONDARY OUTCOMES:
Microbiological quantitative evaluation, bacteria count cfu/ml | 3 months after implant placement
  to assess the presence of the specifical periodontal pathogens, pophyromonas gingivalis all the helaing abutment of the patients in both groups would be taken instad of throuing away and a qualitative analysis will be done on the department of microbiology of the same university.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio caputi, MD, DDS, Principal Investigator — g. d'annunzio chieti-pescara university
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sinjari B, D'Addazio G, De Tullio I, Traini T, Caputi S. Peri-Implant Bone Resorption during Healing Abutment Placement: The Effect of a 0.20% Chlorhexidine Gel vs. Placebo-A Randomized Double Blind Controlled Human Study. Biomed Res Int. 2018 Oct 16;2018:5326340. doi: 10.1155/2018/5326340. eCollection 2018. PMID 30410934